CLINICAL TRIAL: NCT00049816
Title: Aerobic Exercise Intervention for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Kenton R. Kaufman, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AR048768 (NIH); R01AR048768 (NIH); NIAMS-081
Record Dates: First submitted 2002-11-14; First posted 2002-11-15 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Osteoarthritis
Keywords: knee; aerobic exercise; walking; cycling; gait; MRI
MeSH Terms: conditions — Osteoarthritis

ARMS (3):
- 1 (No Intervention): Participants will receive no intervention and will act as the control group.
- 2 (Experimental): Participants will partake in a walking exercise program.
  Interventions: Behavioral: Walking exercise
- 3 (Experimental): Participants will partake in a cycling exercise program.
  Interventions: Behavioral: Cycling Exercise

INTERVENTIONS:
Behavioral: Walking exercise — 30 minutes/day, 3 times/week for 52 weeks
  Arms: 2
Behavioral: Cycling Exercise — 30 minutes/day, 3 times/week for 52 weeks
  Arms: 3

SUMMARY:
This trial will test if walking or bicycling exercise is effective as a non-surgical treatment option for patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Traditional, conservative medical treatment of osteoarthritis has been directed at improving functional status through reducing joint pain and inflammation and maintaining or restoring joint function. Exercise is an adjunct therapy in the clinical management of patients with osteoarthritis of the knee. However, it is not uniformly accepted. The central hypothesis of this work is that the Surgeon General's exercise guidelines can be successfully implemented as an effective nonsurgical option for treatment of patients with early stages of knee osteoarthritis.

Patients with knee osteoarthritis will be randomized into a control group, a walking exercise group, and a stationary cycling exercise group. The individuals in the exercise groups will be required to exercise three times per week for one year using emerging public health recommendations for aerobic exercise in the adult and aging population. Patient outcome will be assessed using objective gait analysis measurements, knee radiographs to quantify joint space narrowing, magnetic resonance imaging, a general health questionnaire (SF-36), a disease/site specific questionnaire (WOMAC), and a visual-analog pain scale. All subjects will be studied at 0 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria

* Current symptoms of chronic (6 months), stable pain and/or stiffness in one or both knees during weight-bearing activities
* Involved joint is primary factor limiting physical or functional activity
* Radiographic signs of mild or moderate arthritis
* Mild joint space narrowing (at least 2mm remaining)

Exclusion Criteria

* Current participation in a regular exercise program
* Existing medical condition that would preclude increased physical activity
* Subjective complaint of instability (giving way)
* Ligamentous instability greater than Grade I
* Knee flexion contracture greater than 15 degrees
* Asymptomatic osteoarthritis of both knees, incapacitating arthritis, or inflammatory arthritis
* Major reconstructive surgery on a lower extremity joint
* Multiple major joint involvement
* Any condition which severely limits local ambulation, such as amputation or stroke
* Gait aids used majority of time for ambulation
* Cannot use step-over-step techniques in either ascending or descending stair conditions
* Not able to undergo MRI scan (e.g., cardiac pacemaker)
* Dementia or inability to give informed consent as determined by a Folstein Mini Mental score greater than 24

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2002-10; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
VAS, SF-36, WOMAC, and Activity Index questionnaires | Week 52
Weight-bearing anterior-posterior (AP) and lateral x-rays of the knee | Week 52
MRI imaging of the knee | Week 52
Measurements of gait during level walking and stair climbing | Week 52

SECONDARY OUTCOMES:
Change in consumption of analgesics, reflecting the level of joint pain | Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Kenton R Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Schmidt JE, Amrami KK, Manduca A, Kaufman KR. Semi-automated digital image analysis of joint space width in knee radiographs. Skeletal Radiol. 2005 Oct;34(10):639-43. doi: 10.1007/s00256-005-0908-9. Epub 2005 May 25. PMID 15915340
- [Background] Grochowski SJ, Amrami KK, Kaufman K. Semi-automated digital image analysis of patellofemoral joint space width from lateral knee radiographs. Skeletal Radiol. 2005 Oct;34(10):644-8. doi: 10.1007/s00256-005-0944-5. Epub 2005 Jul 15. PMID 16021447
- [Background] Koff MF, Amrami KK, Kaufman KR. Clinical evaluation of T2 values of patellar cartilage in patients with osteoarthritis. Osteoarthritis Cartilage. 2007 Feb;15(2):198-204. doi: 10.1016/j.joca.2006.07.007. Epub 2006 Sep 1. PMID 16949313
- [Background] Agnesi F, Amrami KK, Frigo CA, Kaufman KR. Semiautomated digital analysis of knee joint space width using MR images. Skeletal Radiol. 2007 May;36(5):437-44. doi: 10.1007/s00256-006-0245-7. Epub 2007 Jan 23. PMID 17242952
- [Result] Khan FA, Koff MF, Noiseux NO, Bernhardt KA, O'Byrne MM, Larson DR, Amrami KK, Kaufman KR. Effect of local alignment on compartmental patterns of knee osteoarthritis. J Bone Joint Surg Am. 2008 Sep;90(9):1961-9. doi: 10.2106/JBJS.G.00633. PMID 18762657
- [Result] Agnesi F, Amrami KK, Frigo CA, Kaufman KR. Comparison of cartilage thickness with radiologic grade of knee osteoarthritis. Skeletal Radiol. 2008 Jul;37(7):639-43. doi: 10.1007/s00256-008-0483-y. Epub 2008 May 7. PMID 18461323
- [Result] Koff MF, Amrami KK, Felmlee JP, Kaufman KR. Bias of cartilage T2 values related to method of calculation. Magn Reson Imaging. 2008 Nov;26(9):1236-43. doi: 10.1016/j.mri.2008.03.002. Epub 2008 May 7. PMID 18467063